CLINICAL TRIAL: NCT03775252
Title: A Ketogenic Diet Normalizes Interictal Cortical But Not Subcortical Responsivity in Migraineurs
Brief Title: A Ketogenic Diet Acts on Cortical But Not Subcortical Responsivity in Migraineurs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Cherubino DI LORENZO, Principal Investigator, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TrigeMigKeto
Record Dates: First submitted 2018-12-09; First posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Migraine Disorders
Keywords: Ketogenic Diet
MeSH Terms: conditions — Migraine Disorders | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic diet (Experimental): Group of patients treated with ketogenic diet after the first neurophysiological screening.
  Interventions: Dietary Supplement: Ketogenic diet

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — Diet rich in fats and poor in carbohydrate, to induce metabolic ketosis

SUMMARY:
A short ketogenic diet (KD) treatment can prevent migraine attacks and correct excessive cortical response. Here, investigators aim to prove if the KD-related changes of cortical excitability are primarily due to cerebral cortex activity or are modulated by the brainstem.

Through the stimulation of the right supraorbital division of the trigeminal nerve, there will be concurrently interictally recorded the nociceptive blink reflex (nBR) and the pain-related evoked potentials (PREP) in 18 migraineurs patients without aura before and after 1-month on KD, while in metabolic ketosis. nBR and PREP reflect distinct brain structures activation: the brainstem and the cerebral cortex respectively. It will be estimated nBR R2 component area-under-the-curve as well as PREP amplitude habituation as the slope of the linear regression between the 1st and the 2nd block of 5 averaged responses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine
* Kept a headache diary for at least 1 month
* Headache onset before the age of 50

Exclusion Criteria:

* over consumption of acute pain-killers (triptan, analgesic, or ergotamine)
* pregnancy or lactation
* type I diabetes
* serious organic or psychiatric disorders that the investigators judged as having the potential to influence the trial evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Trigeminal neurophysiological changes (amplitude) | one month
  Comparison before and during ketogenic diet of trigeminal neurophysiological features in a population of patients with migraine. In particular, the nociceptive blink reflex (nBR) and the trigeminal pain-related evoked potentials (PREPs) changes of amplitude between the baseline (pre-diet) and during the diet will be used as markers of ketones activity on neural modulation. The unit of measure of the amplitude of neurophysiological evoked responses are the micronVolts (1 volt X 10^-6).
Trigeminal neurophysiological changes (latencies) | one month
  Comparison before and during ketogenic diet of latencies of trigeminal neurophysiological evoked responses in a population of patients with migraine. In particular, the latency of evoked nociceptive blink reflex (nBR) and the trigeminal pain-related evoked potentials (PREPs) changes between the baseline (pre-diet) and during the diet. The unit of measure of the latency of the neurophysiological features are the milliseconds (1 sec X 10^-3).
Trigeminal neurophysiological changes (slope) | one month
  Comparison before and during ketogenic diet of the habituation slope of amplitudes of repeated responses to repetitive trigeminal painful electrical stimuli in a population of patients with migraine. A repetitive stimulus induces repetitive responses from the brainstem and cerebral cortex that physiologically have a decremental trend of amplitudes, also called habituation. On the contrary, in migraineurs, there is a deficit of habituation, i.e. a lack of decremental responses, both in nociceptive blink reflex (nBR) and the trigeminal pain-related evoked potentials (PREPs). The changes induced by ketogenic diet in habituation slope will be measured. The unit of measure of the slope is the radiant degree.

CONTACTS AND LOCATIONS:
Overall Officials: francesco Pierelli, MD, Study Chair — University of Roma La Sapienza
Locations (1):
- Policlinico Umberto I, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
There will be no sharing

REFERENCES:
- [Result] Di Lorenzo C, Coppola G, Bracaglia M, Di Lenola D, Evangelista M, Sirianni G, Rossi P, Di Lorenzo G, Serrao M, Parisi V, Pierelli F. Cortical functional correlates of responsiveness to short-lasting preventive intervention with ketogenic diet in migraine: a multimodal evoked potentials study. J Headache Pain. 2016;17:58. doi: 10.1186/s10194-016-0650-9. Epub 2016 May 31. PMID 27245682
- [Derived] Di Lorenzo C, Coppola G, Bracaglia M, Di Lenola D, Sirianni G, Rossi P, Di Lorenzo G, Parisi V, Serrao M, Cervenka MC, Pierelli F. A ketogenic diet normalizes interictal cortical but not subcortical responsivity in migraineurs. BMC Neurol. 2019 Jun 22;19(1):136. doi: 10.1186/s12883-019-1351-1. PMID 31228957